CLINICAL TRIAL: NCT02296073
Title: The Efficacy and the Safety of Dexmedetomidine Sedation on the PICU Patients-A Randomized, Controlled Study.
Brief Title: The Efficacy and the Safety of Dexmedetomidine Sedation on the Pediatric Intensive Unit(PICU) Patients.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Anhui Provincial Children's Hospital (Other)
Responsible Party: Principal Investigator, Yuanyuan Xu, Anesthesia Department, Anhui Provincial Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PICUDEX2014
Record Dates: First submitted 2014-11-17; First posted 2014-11-20 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Failed Conscious Sedation During Procedure
Keywords: Pediatric intensive care unit; Sedation; Dexmedetomidine; mechanical ventilation
MeSH Terms: interventions — Midazolam; Dexmedetomidine; Fentanyl; Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Midazolam (Experimental): midazolam 3～5μg/kg•min for maintenance of sedation.
  Interventions: Drug: Midazolam; Drug: Fentanyl; Other: assessment
- Dexmedetomidine1 (Experimental): Dexmedetomidine 0.5μg/kg intravenous bump for 15 min，then 0.2～1.4μg/(kg.h) for maintenance of sedation；
  Interventions: Drug: Dexmedetomidine; Drug: Fentanyl; Other: assessment
- Dexmedetomidine2 (Experimental): Dexmedetomidine 0.25μg/kg intravenous bump for 15 min，then 0.2～1.4μg/(kg.h) for maintenance of sedation；
  Interventions: Drug: Dexmedetomidine; Drug: Fentanyl; Other: assessment
- Dexmedetomiding3 (Experimental): Dexmedetomidine 0.2～1.4μg/(kg.h) for maintenance of sedation；
  Interventions: Drug: Dexmedetomidine; Drug: Fentanyl; Other: assessment

INTERVENTIONS:
Drug: Midazolam — midazolam 3～5μg/kg•min for maintenance of sedation.
  Other Names: Liyuexi
  Arms: Midazolam
Drug: Dexmedetomidine — Dexmedetomidine 0.5μg/kg intravenous bump for 15 min，then 0.2～1.4μg/(kg.h) for maintenance of sedation；
  Other Names: Yisi
  Arms: Dexmedetomidine1
Drug: Dexmedetomidine — Dexmedetomidine 0.25μg/kg intravenous bump for 15 min，then 0.2～1.4μg/(kg.h) for maintenance of sedation；
  Other Names: Yisi
  Arms: Dexmedetomidine2
Drug: Dexmedetomidine — Dexmedetomidine 0.2～1.4μg/(kg.h) for maintenance of sedation；
  Other Names: Yisi
  Arms: Dexmedetomiding3
Drug: Fentanyl — Fentanyl 0.5～4 μg/(kg.h) for maintenance of analgesia
  Other Names: Fentai
Other: assessment — Ramsay score for sedation assessment, Facial expression, leg movement, activity, cry, and consolability score (FLACC) for analgesia assessment.

SUMMARY:
To observe the efficacy and safety of dexmedetomidine sedation on the patients admitted to the pediatric intensive care unit after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. written informed consent；
2. pediatric patients admitted to intensive care unit after general anesthesia;
3. expected mechanical ventilation time >6 hours; （4）1 months to 16 years old; -

Exclusion Criteria:

1. congenital heart disease, arrhythmias and heart failure;
2. Alanine transaminase（ALT） and (or) Aspartate aminotransferase（AST） level is more than twice the upper limit of normal;
3. Creatinine and (or) Blood urea nitrogen（BUN） is more than the upper limit of normal;
4. central nervous system disease;
5. spinal analgesia or muscle relaxants is used during PICU;
6. the drug that affects the nerve conduction is used in one month;
7. allergy to the test drug or having other contraindications;
8. participated in other studies 30 days prior to admission of PICU; -

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2014-12; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
percentage of time at target sedation score | up to 24 hours
  assess the sedation level every 2 min using Ramsay score
the number of patients requiring the sedation remedy | up to 24 hours
  the number of patients requiring the sedation remedy during the mechanical ventilation
the dosage of midazolam that need for the sedation remedy | up to 24 hours
  the dosage of midazolam that need for sedation remedy during the mechanical ventilation

SECONDARY OUTCOMES:
change of blood pressure | up to 24 hours.
  the change of blood pressure at 1 min、10 min、20 min、30 min、1 hours、2 hours、3 hours、4 hours、5 hours、6 hours、12 hours、18 hours、24 hours after the sedation drug used.
change of heart rate | up to 24 hours
  the change of heart rate at 1 min、10 min、20 min、30 min、1 hours、2 hours、3 hours、4 hours、5 hours、6 hours、12 hours、18 hours、24 hours after the sedation drug used.
change of respiratory rate | up to 24 hours
  the change of respiratory rate at 1 min、10 min、20 min、30 min、1 hours、2 hours、3 hours、4 hours、5 hours、6 hours、12 hours、18 hours、24 hours after the sedation drug used.
change of blood oxygen saturation | up to 24 hours
  the change of blood oxygen saturation at 1 min、10 min、20 min、30 min、1 hours、2 hours、3 hours、4 hours、5 hours、6 hours、12 hours、18 hours、24 hours after the sedation drug used.
extubation time | up to 24 hours
  time from beginning of study drug used to extubation
change of hepatic function | up to 24 hours
  change of blood ALT、AST level at baseline and 24 hours after the sedation drug used.
change of renal function | up to 24 hours
  change of blood Cr、BUN level at baseline and 24 hours after the sedation drug used.
the dosage of sedation and analgesia drug | up to 24 hours
  the total dosage of sedation and analgesia drug during the sedation and analgesia period
the number of patients requiring fentanyl analgesia in and after 6 hours from study drug used | up to 24 hours
the dosage of fentanyl in and after 6 hours from study drug used | up to 24 hours